CLINICAL TRIAL: NCT01491971
Title: Open-label, Multi-centre, Parallel Group Dose-Escalation Trial Assessing the Pharmacokinetics, Pharmacodynamics, Efficacy and Safety of Intramuscular Injections of Degarelix Administered in 1-Month Dosing Regimens in Patients With Prostate Cancer
Brief Title: Intramuscular Injections of Degarelix Administered in 1-Month Dosing Regimens in Patients With Prostate Cancer
Acronym: IM1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000008
Record Dates: First submitted 2011-11-22; First posted 2011-12-14 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Degarelix - Cohort 1 (Experimental): (gonadotrophin-releasing hormone (GnRH) receptor blocker)
  Interventions: Drug: Degarelix
- Degarelix - Cohort 2 (Experimental): (gonadotrophin-releasing hormone (GnRH) receptor blocker)
  Interventions: Drug: Degarelix
- Degarelix - Cohort 3 (Experimental): (gonadotrophin-releasing hormone (GnRH) receptor blocker)
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix

SUMMARY:
Intramuscular Injections of Degarelix Administered in 1-Month Dosing Regimens in Patients with Prostate Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically confirmed adenocarcinoma of the prostate, for which endocrine therapy is indicated
* Has a current tumour, nodule and metastasis (TNM) staging within 12 weeks prior to treatment start and, if clinically indicated a bone scan
* Has a PSA level meeting one of these criteria:

  1. For treatment-naïve patients: Screening PSA level should be ≥2 ng/mL.
  2. For patients with recurrence after radical prostatectomy: Patients should have a serum PSA increase of ≥0.2 ng/mL from the previous test on two consecutive measurements
  3. For patients with recurrence after radiotherapy or cryotherapy: Patients should have a serum PSA (two measurements) to be >2 ng/mL higher than a previously confirmed PSA nadir
* Has a screening serum testosterone level above the lower limit of normal range in an elderly male population, globally defined as >150 ng/dL
* Has an Eastern Cooperative Oncology Group score of ≤2
* Has a life expectancy of at least one year

Exclusion Criteria:

* Has had previous or is currently under hormonal management of prostate cancer
* Is considered to be a candidate for curative therapy i.e. radical prostatectomy or radiotherapy during the trial period
* Has a history of bilateral orchiectomy, adrenalectomy, or hypophysectomy
* Has a marked baseline prolongation of QT/QTcF interval (e.g. repeated demonstration of a QTcF interval >450 ms)
* Has a history of risk factors for Torsade de Pointes ventricular arrhythmias (e.g. heart failure, hypokalemia, or family history of Long QT Syndrome)
* Has a previous history or presence of another malignancy, other than prostate
* Currently receiving chronic treatment with intramuscular medication injected into the ventrogluteal or dorsogluteal muscle
* Has received an investigational drug within the last 28 days preceding the Screening Visit or longer if considered to possibly influence the outcome of the current trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Plasma degarelix PK profile (blood sample analysis): measured by (Cmax, AUC, Tmax) | Day 0-28 and at Day 112-140
Trough plasma levels (blood sample analysis) | Day 28, 56, 84, 112, 140, 168 and 196
  Actual levels prior to dosing

SECONDARY OUTCOMES:
Proportion of patients with testosterone ≤0.5 ng/mL | From baseline to Day 196
Serum levels of testosterone and PSA | From baseline to Day 196
Percentage change in PSA levels | From baseline to Day 196
Changes in patient-reported injection site pain (VAS scores over time) | At 5 minutes and at 60 minutes after each injection
  Will compare starting dose to maintenance doses
Proportion of patients without clinically significant pain (VAS score of ≤10 mm) | 60 minutes after each dosing injection
Incidence and severity of investigator-evaluated injection site reactions | From baseline to Day 196
Cumulative probabilities of suppressing testosterone to castrate level (≤0.5 ng/mL) by visit | From Day 28 onwards (up to Day 196)
Predictive one-year suppression rate and 95% CI: The cumulative probability of suppressing testosterone to castrate levels (≤0.5 ng/mL) | From Day 28 to Day 364
Incidence of adverse events (AEs) examined by frequency, severity, seriousness and discontinuation from study due to AEs | From baseline to Day 196
Clinically significant changes in laboratory values | From baseline to Day 196
Clinically significant changes in ECGs, vital signs, physical examinations, and body weight | From baseline to Day 196

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (15):
- United States (9):
  - Urology Centers of Alabama, Homewood, Alabama
  - South Orange County Urology Research, Laguna Hills, California
  - San Bernadino Urological Association, San Bernadino, California
  - South Florida Medical Research, Aventura, Florida
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - Carolina Clinical Trials, Concord, North Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Clinic of North Texas, Dallas, Texas
  - Urology San Antonio Research, Pa, San Antonio, Texas
- Canada (6):
  - Pacific Urologic Research, Victoria, British Columbia
  - Euroscope Inc, Barrie, Ontario
  - Bramalea Medical Centre, Brampton, Ontario
  - Urology Associates/Urologic Medical Research, Kitchener, Ontario
  - Office of Dr. Bernard Goldfarb, North Bay, Ontario
  - Urology South Shore Research, Greenfield Park, Quebec